CLINICAL TRIAL: NCT06349993
Title: Digital Intervention for Depression and Anxiety in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adai Technology (Beijing) Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: pd003
Record Dates: First submitted 2024-03-25; First posted 2024-04-05 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Intervention (Experimental)
  Interventions: Behavioral: Digital Intervention
- Health Education (Active Comparator)
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Digital Intervention — game-based digital intervention app
  Arms: Digital Intervention
Behavioral: Health Education — traditional health education app
  Arms: Health Education

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of digital interventions in treating depression and anxiety in adolescents. The main question it aims to answer is: Can digital interventions effectively alleviate symptoms of depression and anxiety in adolescents? The trial will include a comparison group where researchers will compare the effects of the digital intervention to traditional health education methods to assess their relative efficacy.

Participants will be asked to engage with the digital intervention platform for a period of two months.

ELIGIBILITY:
Inclusion Criteria:

* The Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) will be used to assess participants' eligibility based on the diagnostic criteria for depression outlined in the DSM-5(the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition).
* having a HAMD(Hamilton Depression scale) score upon enrollment
* demonstrate normal cognitive function.
* voluntarily agree to participate in the study, and both they and their legal guardians must provide informed consent.

Exclusion Criteria:

* with severe consciousness disorders and a history of psychiatric illness, traumatic brain injury, substance dependence, or acute poisoning
* with concurrent psychiatric disorders (as determined by clinical assessment)
* with concurrent psychiatric disorders (as determined by the assessing clinician)
* at high risk of suicide

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | baseline and immediately after 8-week intervention
  Score Range: 0 (best outcome) to 52 (worst outcome) Higher scores indicate worse depression symptoms.
Hamilton Anxiety Rating Scale | baseline and immediately after 8-week intervention
  Score Range: 0 (best outcome) to 56 (worst outcome) Higher scores indicate more severe anxiety symptoms.

SECONDARY OUTCOMES:
ADHD(attention deficit hyperactivity disorder) Rating Scale-IV | baseline and immediately after 8-week intervention
  Score Range: 0 (best outcome) to 54 (worst outcome) Higher scores indicate more severe ADHD symptoms.
PHQ-9 (Patient Health Questionnaire-9) | baseline and weekly assessments during the treatment period, assessed up to 8 weeks
  PHQ-9 Score Range: 0 (best outcome) to 27 (worst outcome); higher scores indicate more severe depression symptoms.
GAD-7 (Generalized Anxiety Disorder-7) | baseline and weekly assessments during the treatment period, assessed up to 8 weeks
  GAD-7 Score Range: 0 (best outcome) to 21 (worst outcome); higher scores indicate more severe generalized anxiety symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuang, China